CLINICAL TRIAL: NCT05718245
Title: Using Indoor Air Filtration to Reduce PM2.5 Cardiometabolic Effects in At-risk Individuals
Brief Title: HEPA, PM2.5, and Cardiometabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Zhanghua Chen, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: UL2_Study
Record Dates: First submitted 2023-01-24; First posted 2023-02-08 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Air Pollution; Cardiometabolic Health
Keywords: Air pollution; Particulate matter; Air purifier; HEPA filter; Cardiometabolic health

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: A sham filter will be used in the control, to replace HEPA filter in the intervention group. Participants and investigators will be blinded to the intervention type, only specific investigator who will prepare air filter for intervention will be unblinded for the real air filter type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HEPA first and sham (Experimental): This group of participants will be assigned an intervention of HEPA filters with the capacity to reduce PM2.5 levels at their residence for 6 months. After 6-month wash-out period, will be assigned to sham filters for 6 months.
  Interventions: Device: HEPA filter; Device: Sham filter
- Sham first and HEPA (Sham Comparator): This group of participants will be assigned an intervention of sham filters without the capacity to reduce PM2.5 levels at their residence for 6 months. After 6-month wash-out period, will be assigned to HEPA filters for 6 months.
  Interventions: Device: HEPA filter; Device: Sham filter

INTERVENTIONS:
Device: HEPA filter — HEPA filters with the capacity to reduce PM2.5 levels
Device: Sham filter — sham filters without the capacity to reduce PM2.5 levels

SUMMARY:
The goal of this randomized, double-blind, crossover trial is to test the hypothesis that a longer-term indoor HEPA filtration intervention can improve cardiometabolic profiles by reducing indoor PM2.5 exposures in at-risk individuals.

DETAILED DESCRIPTION:
This randomized, double-blind, crossover trial will recruit 52 non-diabetic adults and will investigate potential benefits of HEPA air purifiers on improving cardiometabolic profiles. Participants will be contacted and recruited to the study based on inclusion and exclusion criteria. After consenting, participants will be block randomized to HEPA and control groups for 6-month interventions by sex. After 6-month wash-out period, participants will be switched to the other arm of the intervention. During the trial, project specialists will complete a series of home visits before and after each intervention session to set up air purifiers and indoor and outdoor air pollution monitors, as well as conduct interview to collect questionnaire data, measure body weight and blood pressure, and collect biospecimen. In aim 1, the researcher will assess the effect of a 6-month residential HEPA intervention on changes of type 2 diabetes-related metabolic outcomes in 52 adults. In aim 2, the researchers will examine the association between reduction in indoor PM2.5 exposure brought by the intervention and changes in metabolic outcomes adjusting for ambient PM2.5 exposure. In aim 3, the researchers will explore major pathophysiologic changes pertinent to the cardio-metabolic profile of type 2 diabetes relevance in response to the intervention and changes in PM2.5 exposure.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 and 84 years old;
* Nonsmoker for at least 1 year;
* History of BMI ≥ 25 kg/m2 in the past based on EMR information;
* Either an English or Spanish speaker;
* Live in the Los Angeles County.

Exclusion Criteria:

* History of diabetes (both type 1 and type 2) or degenerative disease of the nervous system (Alzheimer's disease or dementia);
* Currently have active cancer treatment;
* The residential house has already had HEPA filters;
* Participants will move out of the current house in the next 2 years;
* Participants will spend more than one month living outside the primary home;
* Have any health conditions that prohibit collecting health and covariate data and biospecimen;
* The residential houses are not feasible for setting up air purifiers and air pollutants monitors;
* Have high blood glucose from finger stick test (> 200 mg/dL).

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in HOMA-IR | At the baseline and immediately after each of the 6-month interventions
  Difference between baseline and HOMA-IR measured after 6-month intervention
Change in HbA1c | At the baseline and immediately after each of the 6-month interventions
  Difference between baseline and HOMA-IR measured after 6-month intervention

SECONDARY OUTCOMES:
Change in fasting glucose | At the baseline and immediately after each of the 6-month interventions
  Difference between baseline and fasting glucose measured after 6-month intervention
Change in fasting insulin | At the baseline and immediately after each of the 6-month interventions
  Difference between baseline and fasting insulin measured after 6-month intervention
Changes in lipid profiles | At the baseline and immediately after each of the 6-month interventions
  Differences between baseline and LDL, HDL, VLDL, triglycerides, and total cholesterol levels measured after 6-month intervention
Change in blood pressure | At the baseline and immediately after each of the 6-month interventions
  Differences between baseline and systolic and diastolic blood pressure measured after 6-month intervention
Change in continuously monitored glucose level | At the baseline and immediately after 3 months of intervention
  Difference in continuously measured glucose measured using Abbott FreeStyle Libre 2 Pro Continuous Glucose Monitor (CGM) for 2 weeks between baseline and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanghua Chen, PhD, Principal Investigator — University of Southern California; Junfeng Zhang, PhD, Principal Investigator — Duke University
Locations (1):
- Keck School of Medicine, University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No